CLINICAL TRIAL: NCT00142649
Title: Adherence to Weight Loss for Hypertension in African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Purpose: Prevention
Other Study IDs: 250
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Obesity | interventions — Diet; Exercise

INTERVENTIONS:
Behavioral: diet
Behavioral: physical activity

SUMMARY:
To develop a culturally tailored intervention intended to promote adherence to nutrition and physical activity regimens designed to result in weight loss for African American women.

DETAILED DESCRIPTION:
BACKGROUND:

Besides smoking cessation, weight loss and improved nutrition are the most important behavioral changes, which can lead to improved health. Weight loss is also a critically important behavioral recommendation for treating certain illnesses such as hypertension and diabetes; for recovery from stroke or myocardial infarction; and for primary prevention of these conditions as well as certain cancers. Unfortunately, adherence is very poor even with motivated patients. This is a serious issue for all but especially African American women. These diseases affect them disproportionately. They are more likely to be overweight and there is a serious scarcity of culturally appropriate programs available. Also, many of these women receive their care in high demand/low resource clinics so that any program must also be practical and affordable within these constraints.

The study is in response to a Request for Applications issued in January, 2001 on "Overcoming Barriers to Treatment Adherence in Minorities and Persons Living in Poverty."

DESIGN NARRATIVE:

The current research involves studying adherence to recommend changes in behaviors related to nutritional intake and physical activity designed to reduce weight. The investigators will develop and test two versions of a 16-session weight loss program with the content delivered by videotape. They are nearing the end of another study, SisterTalk, for which a culturally appropriate weight control program was designed in partnership with and then delivered to African American women by cable television. Based upon that previous study, they plan to address a number of specific barriers to adherence by designing one version for clinic delivery and another for home delivery. Both approaches, each addressing different adherence issues, will be compared to a Wait List Control Group at 4 and 12 months after beginning the program. The primary outcome measures are adherence to recommended nutritional behaviors and physical activity levels. The program is based upon Social Action Theory and provides the opportunity to study many of that theory's mediating variables and their relationships to specific adherence behaviors. This will include extensive process evaluation procedures.They will also gather a great deal of data concerning the specific barriers and facilitators to adherence to nutrition and physical activity recommendations encountered by low-income African American women who are hypertensive or at high risk for hypertension.

ELIGIBILITY:
No eligibility criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lasater — Brown University